CLINICAL TRIAL: NCT06936540
Title: The Effect of Training on Surgical Environments Provided With Virtual Tour Before Orthopedic Surgical Intervention on Patients' Anxiety and Satisfaction Level
Brief Title: The Effect of Virtual Tour Training Before Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seda Baydemir, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IUC-SN-SB-01
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Satisfaction
Keywords: Anxiety; Satisfaction; Virtual Reality; Orthopedic Surgical Procedures
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: The study was planned as an open-label, randomized, controlled, parallel group interventional study. Participants will be randomly assigned to either the intervention group or the control group. The intervention group will be trained by the researcher with a virtual tour material about surgical environments via a tablet computer. The control group will not receive any intervention other than verbal training in the routine of the organization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): The intervention group will be trained by the researcher with a virtual tour material about surgical environments via a tablet computer.
  Interventions: Other: Virtual Tour
- Control group (Other): The control group will not receive any intervention other than verbal training in the routine of the organization.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: Virtual Tour — The intervention group will be trained by the researcher with a virtual tour material about surgical environments via a tablet computer.
  Arms: Intervention group
Other: No Interventions — The control group will not receive any intervention other than verbal training in the routine of the organization.
  Arms: Control group

SUMMARY:
The purpose of the study is to determine the effect of training on surgical environments provided with virtual tour before orthopedic surgical ıntervention on patients' anxiety and satisfaction level.

DETAILED DESCRIPTION:
Although preoperative anxiety is accepted as a normal patient response, severe anxiety can lead to a number of negative physiological, emotional and cognitive consequences for patients and ultimately to prolonged hospitalization. If anxiety is not managed effectively in the preoperative period, recovery time is prolonged and the risk of anesthesia and surgery-related complications increases. Moreover, it can lead to respiratory distress and cardiac problems. It causes life threats by increasing the risk of bleeding with deterioration in hemodynamic parameters and negatively affects surgical outcomes and patient satisfaction. For all these reasons, this study was designed to contribute to the management of anxiety, which is seen as a problem that needs to be addressed in surgical nursing.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Being literate
* No comprehension and perception problems
* No hearing and vision problems
* Not being under psychiatric treatment
* No surgical experience
* To undergo elective orthopedic surgery in the operating room
* Acceptance to participate in the research

Exclusion Criteria:

* To undergo emergency orthopedic surgery
* Wishing to leave at any stage of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-04-12 (Actual); Primary Completion 2025-10-12 (Actual); Study Completion 2025-10-12 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI): Pre-test and post-test differences of anxiety levels | From immediately before preoperative training to immediately after preoperative training (on the day before surgery).
  The State-Trait Anxiety Inventory (STAI) is accepted as the the gold standard to determine the level of anxiety. The validity and reliability of the STAI in Turkey was conducted by Oner and Le Compte. The STAI can be administered to individuals over the age of 14 and there is no time limit for answering. It includes two separate scales of twenty items each (ie, the State Anxiety Scale (STAI-S) and the Trait Anxiety Scale (STAI-T). STAI-S and STAI-T scores are calculated separately. The total score obtained from the scales varies between 20 and 80, and a high score indicates a high level of anxiety.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for Satisfaction: Pre-test and post-test differences of satisfaction levels | From immediately before preoperative training to immediately after preoperative training (on the day before surgery).
  The satisfaction form, created by the researcher using the Visual Analog Scale (VAS), includes a scale for patients to rate their satisfaction. Scoring is between 0 and 10 points (0 to 10 inclusive). A high score indicates a high level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Baydemir, PhD-candidate, Principal Investigator — Istanbul University-Cerrahpasa Institute of Graduate Studies
Locations (1):
- Istanbul University-Cerrahpasa Institute of Graduate Studies, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No